CLINICAL TRIAL: NCT07213973
Title: A Phase 2, Open-Label Study to Evaluate the Safety, Pharmacokinetics, and Efficacy of Povorcitinib in Adolescents With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Pharmacokinetics, Safety, and Efficacy of Povorcitinib in Adolescent Participants With Moderate to Severe Hidradenitis Suppurativa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB054707-211
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: Hidradenitis Suppurativa; HS; INCB054707; Povorcitinib; Acne inversa; Hidradenitis
MeSH Terms: conditions — Hidradenitis Suppurativa; Hidradenitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Povorcitinib Dose A (Experimental): Participants will receive povorcitinib dose A for 54 weeks.
  Interventions: Drug: Povorcitinib
- Povorcitinib Dose B (Experimental): Participants will receive povorcitinib dose B for 54 weeks.
  Interventions: Drug: Povorcitinib

INTERVENTIONS:
Drug: Povorcitinib — Oral; Tablet
  Other Names: INCB054707

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety, and efficacy of povorcitinib in adolescent participants with moderate to severe hidradenitis suppurativa over a 54-week open-label treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 12 to < 18 years at the time of informed consent/assent signing.
* Body weight ≥ 30 kg at both screening and baseline visits.
* Diagnosis of moderate to severe HS for at least 3 months prior to the screening visit.
* Total abscess and inflammatory nodule count of at least 5 at both the screening and baseline visits.
* HS lesions corresponding to refined Hurley Stage IB, IC, IIB, IIC, or III at both the screening and baseline visits.
* Documented history of inadequate response to at least a 3-month course of at least 1 conventional systemic therapy (oral antibiotic or biologic drug) for HS (or demonstrated intolerance to, or have a contraindication to, a conventional systemic therapy for treatment of their HS).
* Agreement to use contraception.
* Willing and able to comply with the study protocol and procedures.
* Further inclusion criteria apply.

Exclusion Criteria:

* Presence of > 20 draining tunnels (fistulas) at either the screening or baseline visit.
* Women who are pregnant (or who are considering pregnancy) or breastfeeding.
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q-wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
* Laboratory values outside of the protocol-defined ranges.
* Further exclusion criteria apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2028-03-25 (Estimated); Study Completion 2028-03-25 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with Treatment-Emergent Adverse Events (TEAEs) | Baseline through Week 54
  TEAE is defined as any AE either reported for the first time or worsening of a pre-existing event after the first dose of study drug up to 30 days after the last dose of study drug.
Apparent clearance | Up to Week 24
Apparent volume of distribution | Up to Week 24
Apparent oral absorption rate constant | Up to Week 24
Absorption lag time | Up to Week 24
Maximum plasma drug concentration at steady state | Up to Week 24
Average plasma drug concentration at steady state | Up to Week 24
Plasma concentration at steady state for the dosing interval | Up to Week 24
Time to maximum plasma concentration at steady state | Up to Week 24
Terminal half-life | Up to Week 24

SECONDARY OUTCOMES:
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 50 (HiSCR50) | 54 weeks
  HiSCR50 is defined as at least a 50% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) | 54 weeks
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and inflammatory nodule count, with no increase from baseline in abscess or draining tunnel count.
Mean change from baseline in abscess count at each visit | 54 weeks
  Defined as mean change of abscess count relative to baseline.
Mean percentage change from baseline in abscess count at each visit | 54 weeks
  Defined as mean percentage change from baseline in abscess count.
Mean change from baseline in inflammatory nodule count at each visit | 54 weeks
  Defined as mean change of inflammatory nodule count relative to baseline.
Mean percentage change from baseline in inflammatory nodule count at each visit | 54 weeks
  Defined as mean percentage change from baseline in inflammatory nodule count.
Mean change from baseline in draining tunnel count at each visit | 54 weeks
  Defined as mean change of draining tunnel count relative to baseline.
Mean percentage change from baseline in draining tunnel count at each visit | 54 weeks
  Defined as mean percentage change from baseline in draining tunnel count.
Proportion of participants who achieve Skin Pain Numeric Rating Scale (NRS)30 among participants with baseline Skin Pain NRS score ≥ 3 | 54 weeks
  Defined as participants with a Skin Pain NRS score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Proportion of participants with a ≥ 3-point decrease in Skin Pain NRS score among participants with baseline Skin Pain NRS score ≥ 3 | 54 weeks
  Participants with a Skin Pain score of at least 3 at baseline and who experience at least a 3-point decrease in Skin Pain score.
Change from baseline in Children's Dermatology Life Quality Index (CDLQI) score at each visit | 54 weeks
  The CDLQI is a simple, 10-question validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days, across symptoms and feelings, leisure, school or holidays, personal relationships, sleep, and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical Monitor, Study Director — Incyte Corporation
Locations (30):
- United States (25):
  - University of Alabama At Birmingham, Birmingham, Alabama
  - Medical Dermatology Specialists Phoenix, Phoenix, Arizona
  - Saguaro Dermatology, Phoenix, Arizona
  - Rady Children'S Hospital-San Diego, San Diego, California
  - Uconn Health, Farmington, Connecticut
  - University of Miami Miller School of Medicine, Miami, Florida
  - Skin Research of South Florida, Llc, Miami, Florida
  - Trueblue Clinical Research, Tampa, Florida
  - Marietta Dermatology the Skin Cancer Center Marietta, Marietta, Georgia
  - Advanced Medical Research Pc, Sandy Springs, Georgia
  - Endeavor Health Medical Group, Skokie, Illinois
  - Dermatology Skin Cancer Center Leawood, Leawood, Kansas
  - Equity Medical, Bowling Green, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Boston Childrens Hospital, Boston, Massachusetts
  - Oakland Hills Dermatology Pc, Auburn Hills, Michigan
  - Wayne State University Physician Group Dermatology, Detroit, Michigan
  - Revival Research Institute, Llc Troy, Troy, Michigan
  - Washington University, St Louis, Missouri
  - Boeson Research Missoula 2825 Fort Missoula Rd, Missoula, Montana
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - Geisinger Medical Center, Danville, Pennsylvania
  - Bellaire Dermatology Associates Bda, Bellaire, Texas
  - Texas Dermatology Research Center, Dallas, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
- Canada (5):
  - Beacon Dermatology, Calgary, Alberta
  - Dermcare Clinic, Mississauga, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - The Hospital For Sick Children, Toronto, Ontario
  - Skincare Studio Dermatology Centre, St. John's

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Pharmacokinetics, Safety, and Efficacy of Povorcitinib in Adolescent Participants With Moderate to Severe Hidradenitis Suppurativa — https://incyteclinicaltrials.com/studies/nct07213973